CLINICAL TRIAL: NCT02224820
Title: A Phase II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of Intravenous IdeS After Administration of Ascending Doses in Chronic Kidney Disease Patients
Brief Title: Phase II Study, Evaluation of Safety and Efficacy of IdeS in Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-HMedIdeS-02; 2013-005417-13 (EudraCT Number)
Record Dates: First submitted 2014-08-15; First posted 2014-08-25 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Chronic Kidney Disease
Keywords: transplantation; sensitised patients; HLA-antibodies
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intravenous IdeS (Experimental): One or two doses of IdeS in ascending doses
  Interventions: Biological: IdeS

INTERVENTIONS:
Biological: IdeS — Doses are administered in ascending doses

SUMMARY:
IdeS is an immunoglobulin g (IgG) cleaving enzyme. It will given to patients with donor specific antibodies to reduce the antibody load and thus enable kidney transplantation. IdeS antibody reducing efficacy and its safety will be studied.

DETAILED DESCRIPTION:
Study 13-HMedIdeS-02 (EudraCT no. 2013-005417-13) is a single centre, single arm, dose finding, Phase II study in sensitized CKD patients assessing safety, tolerability, pharmacokinetics (PK) and efficacy of HMED-IdeS without intent to transplantation. However, patients are not removed from the transplant waitlist during the study. Included patients has a panel reactive antibody [PRA] >70% (n=7).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic kidney disease and in dialysis with identified antibodies against at least two HLA antigens of which at least one is 3000 MFI or more as measured by SAB assay on at least two occasions.

Exclusion Criteria:

* Prior malignancy within 2 years excluding adequately treated basal cell or squamous cell skin cancer, cervical carcinoma in situ and prostate cancer Gleason <6 and prostate-specific antigen (PSA) <10 ng/mL.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus (HIV
* Clinical signs of ongoing infectious disease.
* Severe other conditions requiring treatment and close monitoring, e.g. cardiac failure > New York Heart Association (NYHA) grade 3, unstable coronary disease or oxygen dependent chronic obstructive pulmonary disease (COPD)
* History of any other clinically significant disease or disorder which, in the opinion of the investigator, may either put the patient at increased risk because of participation in the study, or influence the results or the patient's ability to participate in the study
* Hypogammaglobulinemia defined as any values of P-total IgG less than 3 g/L
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to IdeS (e. g streptokinase and/or staphylokinase)
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical study that included drug treatment within 4 months of the first administration of investigational product in this study. Patients consented and screened but not dosed in previous studies are not excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Lorant, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Dept. of Transplant Surgery, Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bockermann R, Jarnum S, Runstrom A, Lorant T, Winstedt L, Palmqvist N, Kjellman C. Imlifidase-generated Single-cleaved IgG: Implications for Transplantation. Transplantation. 2022 Jul 1;106(7):1485-1496. doi: 10.1097/TP.0000000000004031. Epub 2021 Dec 27. PMID 34966107
- [Derived] Lorant T, Bengtsson M, Eich T, Eriksson BM, Winstedt L, Jarnum S, Stenberg Y, Robertson AK, Mosen K, Bjorck L, Backman L, Larsson E, Wood K, Tufveson G, Kjellman C. Safety, immunogenicity, pharmacokinetics, and efficacy of degradation of anti-HLA antibodies by IdeS (imlifidase) in chronic kidney disease patients. Am J Transplant. 2018 Nov;18(11):2752-2762. doi: 10.1111/ajt.14733. Epub 2018 Apr 17. PMID 29561066
- [Derived] Jordan SC, Lorant T, Choi J, Kjellman C, Winstedt L, Bengtsson M, Zhang X, Eich T, Toyoda M, Eriksson BM, Ge S, Peng A, Jarnum S, Wood KJ, Lundgren T, Wennberg L, Backman L, Larsson E, Villicana R, Kahwaji J, Louie S, Kang A, Haas M, Nast C, Vo A, Tufveson G. IgG Endopeptidase in Highly Sensitized Patients Undergoing Transplantation. N Engl J Med. 2017 Aug 3;377(5):442-453. doi: 10.1056/NEJMoa1612567. PMID 28767349

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed at a medical clinic, the Department of Transplantat Surgery, Uppsala, SE between 10 Jun 2014 and 13 Feb 2015. The patients had chronic kidney disease, were in dialysis and on the waiting list for transplantation. (Transplantation was not part of the protocol).
Pre-assignment Details: In total, 10 patients were assessed for eligibility. One patient declined to participate and one patient was not available for recieving information about the study. Eight patients were enrolled and started treatment.
Period: Overall Study
Arm/Group | Intravenous IdeS
Started | 8
Completed | 8 (One patient did not receive full dose)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 0ne patient interrupted treatment.
Groups:
- Intravenous IdeS: One or two doses of IdeS in ascending doses
  IdeS
Arm/Group | Intravenous IdeS
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (11.9)
Gender [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Weight (kg) [Mean (Standard Deviation); unit: kg] | 74.5 (14.5)
BMI [Mean (Standard Deviation); unit: kg/mg^2] | 25.1 (4.5)
Height [Mean (Standard Deviation); unit: cm] | 172.3 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy
Description: Efficacy was defined as the IdeS dosing scheme in the majority of the patients resulting in human leucocyte antigen (HLA) antibody levels which are acceptable for transplantation, measured as mean fluorescent intensity (MFI) of less than 1100, within 24 hours from dosing. MFI was determined by single antigen bead (SAB) assay and detection of complement fixating ability (CIq Screen) in serum.
Time Frame: 24 hours
Measure: Mean (Inter-Quartile Range); unit: MFI
Arm/Group | Intravenous IdeS
Number analyzed (Participants) | 8
MFI | 372 [83 to 978]

2. Secondary Outcome: Safety
Description: Adverse events (all clinical laboratory tests, vital signs and ECG jugded as clinically significant were reported as AEs)
Time Frame: 9 weeks
Measure: Number; unit: Adverse events
Arm/Group | Intravenous IdeS
Number analyzed (Participants) | 8
Adverse events | 76

3. Secondary Outcome: Pharmacodynamics
Description: IgG cleavage and regeneration measured by ELISA
Time Frame: Up to day 64
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Intravenous IdeS
Number analyzed (Participants) | 8
µg/mL | 30 (3)

4. Secondary Outcome: Immunogenicity
Description: Presence of Anti-Drug Antibodies formation in serum throughout a 64 day period
Time Frame: Up to 64 days
Measure: Number; unit: participants
Arm/Group | Intravenous IdeS
Number analyzed (Participants) | 8
participants | 8

5. Secondary Outcome: Pharmacokinetics
Description: IdeS T1/2 in alpha phase. One patient who interrupted dose was excluded.
Time Frame: Up to 21 days
Measure: Mean (Inter-Quartile Range); unit: h
Arm/Group | Intravenous IdeS
Number analyzed (Participants) | 7
h | 5 [2 to 11]

ADVERSE EVENTS:
Time Frame: From the time of admission until last visit, 64 days after treatment.
Arm/Group | Intravenous IdeS
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous IdeS (N=8)
Pneumonia (Infections and infestations) | 2 (2)
Suspected upper respiratory infection (Infections and infestations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased mucos production (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous IdeS (N=8)
Nasopharyngitis (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Herpes simplex infection (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferas increased (Investigations) | 2 (2)
Aspartate aminotransferas increased (Investigations) | 2 (2)
Blood phosphorus increased (Investigations) | 1 (1)
C-reactive proteine increased (Investigations) | 1 (1)
Donor specific antibody present (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Dyspesia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Infusion site pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Feeling cold (General disorders) | 1 (1)
Feeling hot (General disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Leucocytosis (Blood and lymphatic system disorders) | 2 (2)
Leucopenia (Blood and lymphatic system disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1)
Dysgeuisa (Nervous system disorders) | 1 (1)
Flushing (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Scleral haemorrage (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 1 (1) — Dose was interrupted for this patient due to infusion reaction.The pat was transplanted (not defined as SAE in protocol) 4 days after dosing. Pat remained in the study for safety follow-up. A number of AEs related to the transplantation are reported.
Haematuria (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No